CLINICAL TRIAL: NCT01993810
Title: Phase III Randomized Trial Comparing Overall Survival After Photon Versus Proton Chemoradiotherapy for Inoperable Stage II-IIIB NSCLC
Brief Title: Comparing Photon Therapy To Proton Therapy To Treat Patients With Lung Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 1308; NCI-2013-01850 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RTOG 1308; RTOG-1308 (Other: NRG Oncology); RTOG-1308 (Other: CTEP); U10CA180868 (NIH); U10CA021661 (NIH)
Record Dates: First submitted 2013-11-12; First posted 2013-11-25 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Stage II Non-Small Cell Lung Cancer AJCC v7; Stage IIA Non-Small Cell Lung Carcinoma AJCC v7; Stage IIB Non-Small Cell Lung Carcinoma AJCC v7; Stage III Non-Small Cell Lung Cancer AJCC v7; Stage IIIA Non-Small Cell Lung Cancer AJCC v7; Stage IIIB Non-Small Cell Lung Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; durvalumab; Immunoglobulin G; Disulfides; Etoposide; Paclitaxel; Taxes; Pemetrexed; Proton Therapy; Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (photon beam radiation therapy and chemotherapy) (Active Comparator): Patients undergo photon beam radiation therapy 5 days per week for a total of 35 fractions and receive either paclitaxel* IV over 1 hour and carboplatin* IV weekly during radiation therapy or etoposide IV on days 1-5 and 29-33 and cisplatin IV on days 1, 8, 29, and 36. Patients with non-squamous cell cancer may receive pemetrexed IV and carboplatin IV on every 21 days. Patients who receive paclitaxel and carboplatin must complete 2 courses of consolidation therapy.
  CONSOLIDATION THERAPY: Beginning 3-6 weeks after chemoradiotherapy, patients receive either paclitaxel IV over 3 hours and carboplatin IV on day 1 or durvalumab IV every 2 weeks. Treatment repeats every 21 days for 2 courses or every 2 weeks for up to 12 months for durvalumab in the absence of disease progression or unacceptable toxicity. Patients with non-squamous cell carcinoma may receive durvalumab or pemetrexed IV and carboplatin IV on day 1 every 21 days for up to 4 courses.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Biological: Durvalumab; Drug: Etoposide; Drug: Paclitaxel; Drug: Pemetrexed Disodium; Radiation: Photon Beam Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (proton beam radiation therapy and chemotherapy) (Experimental): Patients undergo proton beam radiation therapy 5 days per week for a total of 35 fractions and receive either paclitaxel* and carboplatin*, etoposide and cisplatin, or pemetrexed and carboplatin (for non-squamous cell cancer patients only) as in Arm I. Patients who receive paclitaxel and carboplatin must complete 2 courses of consolidation therapy.
  CONSOLIDATION THERAPY: Beginning 3-6 weeks after chemoradiotherapy, patients receive either paclitaxel IV over 3 hours and carboplatin IV on day 1 or durvalumab IV every 2 weeks. Treatment repeats every 21 days for 2 courses or every 2 weeks for up to 12 months for durvalumab in the absence of disease progression or unacceptable toxicity. Patients with non-squamous cell carcinoma may receive durvalumab or pemetrexed IV and carboplatin IV on day 1 every 21 days for up to 4 courses.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Biological: Durvalumab; Drug: Etoposide; Drug: Paclitaxel; Drug: Pemetrexed Disodium; Radiation: Proton Beam Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Drug: Pemetrexed Disodium — Given IV
  Other Names: Alimta; LY231514; N-[4-[2-(2-Amino-4,7-dihydro-4-oxo-1H-pyrrolo[2,3-d]pyrimidin-5-yl)ethyl]benzoyl]-L-glutamic Acid Disodium Salt
Radiation: Photon Beam Radiation Therapy — Undergo photon beam radiation therapy
  Arms: Arm I (photon beam radiation therapy and chemotherapy)
Radiation: Proton Beam Radiation Therapy — Undergo proton beam radiation therapy
  Other Names: PBRT; Proton Radiation Therapy
  Arms: Arm II (proton beam radiation therapy and chemotherapy)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase III trial studies proton chemoradiotherapy to see how well it works compared to photon chemoradiotherapy in treating patients with stage II-IIIB non-small cell lung cancer that cannot be removed by surgery. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor, such as photon or proton beam radiation therapy, may kill more tumor cells and cause less damage to normal tissue. Drugs used in chemotherapy, such as paclitaxel, carboplatin, etoposide, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether proton chemoradiotherapy is more effective than photon chemoradiotherapy in treating non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the overall survival (OS) in patients with stage II-IIIB non-small cell lung cancer (NSCLC) after image guided, motion-managed photon radiotherapy (Arm 1) or after image guided, motion-managed proton radiotherapy (Arm 2) both given with concurrent platinum- based chemotherapy.

II. To compare the cardiac toxicity and lymphocyte reduction (lymphopenia) definitely, probably, or possibly related to treatment between the 2 arms.

SECONDARY OBJECTIVES:

I. To compare 2-year progression-free survival (PFS) between the 2 arms. II. To compare the development of grade 3 or higher adverse events not included above that are definitely, probably, or possibly related to treatment.

III. To compare differences between the two arms in quality of life (QOL) based primarily on the development of shortness of breath at 6 months and secondarily on the development of sore throat at the end of chemoradiotherapy (chemoRT) (as measured by the lung cancer module of the MD Anderson Symptom Inventory [MDASI-Lung]), as well as breathing related functioning impairments as measured by the Shortness Breath Questionnaire [SOBQ].

IV. To compare cost-effectiveness outcomes between the 2 arms. V. To compare pulmonary function changes by treatment arms and response. VI. To explore the most appropriate and clinically relevant technological parameters to ensure quality and effectiveness throughout radiation therapy processes, including imaging, simulation, patient immobilization, target and critical structure definition, treatment planning, image guidance and delivery.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo photon beam radiation therapy 5 days per week for a total of 35 fractions and receive either paclitaxel* intravenously (IV) over 1 hour and carboplatin* IV weekly during radiation therapy or etoposide IV on days 1-5 and 29-33 and cisplatin IV on days 1, 8, 29, and 36. Patients with non-squamous cell cancera may receive pemetrexed IV and carboplatin IV on every 21 days.

ARM II: Patients undergo proton beam radiation therapy 5 days per week for a total of 35 fractions and receive either paclitaxel* and carboplatin*, etoposide and cisplatin, or pemetrexed and carboplatin (for non-squamous cell cancer patients only) as in Arm I.

*In both arms, patients who receive paclitaxel and carboplatin must complete 2 courses of consolidation therapy.

CONSOLIDATION THERAPY: Beginning 3-6 weeks after chemoradiotherapy, patients receive either paclitaxel IV over 3 hours and carboplatin IV on day 1 or durvalumab IV every 2 weeks. Treatment repeats every 21 days for 2 courses or every 2 weeks for up to 12 months for durvalumab in the absence of disease progression or unacceptable toxicity. Patients with non-squamous cell carcinoma may receive durvalumab or pemetrexed IV and carboplatin IV on day 1 every 21 days for up to 4 courses.

After completion of study treatment, patients are followed up at 4-8 weeks, every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of non-small cell lung cancer
* Clinical American Joint Committee on Cancer (AJCC) (AJCC, 7th ed.) II, IIIA or IIIB (with non-operable disease; non-operable disease will be determined by a multi-disciplinary treatment team within 60 days prior to registration; note: for patients who are clearly nonresectable, the case can be determined by the treating radiation oncologist and/or a medical oncologist or pulmonologist

  * Patients who present with N2 or N3 disease and an undetectable NSCLC primary tumor are eligible
  * Patients who refuse surgery are eligible
  * Patients who develop local recurrence after surgery and rendered candidate for definitive concurrent chemoradiation are also eligible
  * Patients who have received systemic treatment (up to 4 cycles of induction chemotherapy, or up to 6 months of targeted therapy) are eligible
* Appropriate stage for protocol entry, including no distant metastases, based upon the following minimum diagnostic workup:

  * History/physical examination within 30 days prior to registration including resting heart rate;
  * Fludeoxyglucose F 18 (FDG)-positron emission tomography (PET)/computed tomography (CT) scan for staging within 60 days prior to registration
  * Magnetic resonance imaging (MRI) scan with contrast of the brain (preferred) or CT scan of the brain with contrast within 60 days prior to registration;
  * Forced expiratory volume in one second (FEV1) >= 0.8 liter or >= 35% predicted with or without bronchodilator within 90 days prior to registration;

    * Patients who meet the criterion above without oxygen (O2), but who need acute (started within 10 days prior to registration) supplemental oxygen due to tumor-caused obstruction/hypoxia are eligible, provided the amount of the O2 needed has been stable
* Zubrod performance status 0-1 within 30 days prior to registration
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3 obtained within 30 days prior to registration
* Platelets >= 100,000 cells/mm^3 obtained within 30 days prior to registration
* Hemoglobin >= 9.0 g/dl (note: the use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 9.0 g/dl is acceptable), obtained within 30 days prior to registration
* Serum glutamic oxaloacetic transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) within 30 days prior to registration

  * It is highly recommended but not required that SGOT or SGPT be =< 1.5 upper limit of normal
* Total bilirubin =< 1.5 within 30 days prior to registration

  * It is highly recommended but not required that total bilirubin be =< 1.5 upper limit of normal
* Serum creatinine < 1.5 mg/dL or calculated creatinine clearance >= 50 mL/min within 30 days prior to registration estimated by the Cockcroft-Gault formula
* Peripheral neuropathy =< grade 1 at the time of registration
* Patients with non-malignant pleural effusion are eligible

  * If a pleural effusion is present, the following criteria must be met to exclude malignant involvement:

    * When pleural fluid is visible on both the CT scan and on a chest x-ray, a pleuracentesis is required to confirm that the pleural fluid is cytologically negative
    * Exudative pleural effusions are excluded, regardless of cytology
    * Effusions that are minimal (i.e, not visible on chest x-ray) that are too small to safely tap are eligible
* Patients must have measurable or evaluable disease
* Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to registration
* Women of childbearing potential and male participants must practice adequate contraception
* Patient must provide study-specific informed consent prior to study entry

Exclusion Criteria:

* Prior invasive malignancy unless disease free for a minimum of 3 years; however, skin cancer and in situ carcinomas of the breast, oral cavity, cervix, and other organs and are permissible
* Patients with prior history of either small cell lung cancer or NSCLC regardless of the treatment received, other than patients who have recurrent disease following resection
* Prior systemic chemotherapy for the study cancer, if more than 4 cycles of induction chemotherapy or more than 6 months of targeted therapy; note that prior chemotherapy for a different cancer is allowable
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months;
  * Transmural myocardial infarction within the last 6 months;
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness other than the diagnosed lung cancer requiring hospitalization or precluding study therapy within 30 days before registration;
  * Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that human immunodeficiency virus (HIV) testing is not required for entry into this protocol
* Unintentional weight loss > 10% within 30 days prior to registration
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2014-02-03 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From registration until death or last follow-up; analysis occurs after 390 deaths have been reported
  The time from study registration until death or last follow-up

SECONDARY OUTCOMES:
Progression-free survival | From registration to date of local failure, regional failure, distant failure, death from any cause, or until last follow-up. Analysis occurs after 390 deaths have been reported.
  The time from study registration until the first occurrence of local, regional, or distant progression, or death from any cause, or until last follow-up
Adverse events | From start of treatment to end of follow-up
  Incidence of treatment-related grade 3-5 adverse events, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Zhongxing Liao, Principal Investigator — NRG Oncology
Locations (30):
- United States (30):
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Upper Chesapeake Medical Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - Tate Cancer Center, Glen Burnie, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - ProCure Proton Therapy Center-Somerset, Somerset, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - West Chester Hospital, West Chester, Ohio
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Tennessee Cancer Specialists-Dowell Springs, Knoxville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson Regional Care Center-Katy, Houston, Texas
  - MD Anderson Regional Care Center-Bay Area, Nassau Bay, Texas
  - MD Anderson Regional Care Center-Sugar Land, Sugar Land, Texas
  - MD Anderson Regional Care Center-The Woodlands, The Woodlands, Texas
  - ProCure Proton Therapy Center-Seattle, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Ramella S, D'Angelillo RM. Proton beam or photon beam radiotherapy in the treatment of non-small-cell lung cancer. Lancet Oncol. 2020 Jul;21(7):873-875. doi: 10.1016/S1470-2045(20)30246-1. No abstract available. PMID 32615102